CLINICAL TRIAL: NCT05817084
Title: Outcomes of Anterior Cruciate Ligament Reconstruction With and Without High Tibial Osteotomy in Knees With Varus Malalignment. Comparative Study
Brief Title: Patients With Acl Injury and Varus Knee Will Undergo Acl Reconstruction Alone, or Combined With High Tibial Osteotomy in the Same Session.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mostafa Hassanein, Msc (Other)
Responsible Party: Sponsor-Investigator, Mostafa Hassanein, Msc, principal investigator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD80/2022
Record Dates: First submitted 2023-03-10; First posted 2023-04-18 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: ACL - Anterior Cruciate Ligament Deficiency; Varus Deformity of Tibia (Disorder); ACL Injury; Knee Deformity
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12 patients with varus knee malalignment and acl deficiency under went acl reconstruction and hto (Active Comparator): anterior cruciate ligament reconstruction and medial opening wedge high tibial osteotomy in the same session
  Interventions: Procedure: medial opening wedge high tibial osteotomy; Procedure: anterior cruciate ligament reconstruction
- 12 patients with varus knee malalignment and acl deficiency underwent acl reconstruction (Active Comparator): anterior cruciate ligament reconstruction alone.
  Interventions: Procedure: anterior cruciate ligament reconstruction

INTERVENTIONS:
Procedure: medial opening wedge high tibial osteotomy — medial opening wedge valgus high tibial osteotomy
  Arms: 12 patients with varus knee malalignment and acl deficiency under went acl reconstruction and hto
Procedure: anterior cruciate ligament reconstruction — anterior cruciate ligament reconstruction

SUMMARY:
The purpose of this study is to compare the results of single-stage anterior cruciate ligament reconstruction combined with high tibial osteotomy and anterior cruciate ligament reconstruction alone in knees with varus malalignment and anterior cruciate ligament deficiency. Evaluation will be clinically, radiologically and time needed to return to pre injury activity level. Our Hypothesis: Simultaneous anterior cruciate ligament reconstruction and high tibial osteotomy provides good functional scores, low rate of graft failure and early return to pre injury activity level with minimal added morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 50.
* Knee varus malalignment 7-10°.
* ACL injury with clinical anterior instability confirmed by MRI.

Exclusion Criteria:

* Osteoarthritis (Kellgren-Lawrence grade IV).
* Inflammatory joint disease.
* Knee flexion < 120°
* Knee fixed flexion deformity > 10°.
* BMI >30
* Any ligamentous or meniscal knee injury other than ACL injury.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Lysholm knee score | 1 month post operative
  knee score from 0 to 100 where a higher score means better outcome.
Lysholm knee score | 3 month post operative
  knee score from 0 to 100 where a higher score means better outcome.
Lysholm knee score | 6 month post operative
  knee score from 0 to 100 where a higher score means better outcome.
Tegner activity level | 1 month post operative
  activity level from 0 to 11 where 11 means highest level
Tegner activity level | 3 months post operative
  activity level from 0 to 11 where 11 means highest level
Tegner activity level | 6 months post operative
  activity level from 0 to 11 where 11 means highest level
Return to pre injury level | through study completion, an average of 7 months
  time needed by the patient in months post operative to return to pre injury activity level

SECONDARY OUTCOMES:
knee range of motion | pre operative, 1 month, 3months, and 6 months post operative
  measure knee range of motion in degrees "flexion and extension"
knee stability | pre operative, 1 month, 3months, and 6 months post operative
  Lachman knee stability test

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No